CLINICAL TRIAL: NCT05210270
Title: Phase 1/2 Trial Evaluating the Effectiveness and Safety of Dose-adapted HYpofractionated Pelvic Radiotherapy for Advanced Cervical Cancers INeligible for ChemoTherapy
Brief Title: HYpofractionated Pelvic Radiotherapy for Advanced Cervical Cancers INeligible for ChemoTherapy
Acronym: HYACINCT
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Santo Tomas Hospital, Philippines (Other)
Collaborators: Philippine Council for Health Research & Development (Other Government)
Responsible Party: Principal Investigator, Warren Bacorro, Doctor, University of Santo Tomas Hospital, Philippines
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USTH-BCI-RO-2022-01; REC-2021-08-104-CT (Other: University of Santo Tomas Hospital)
Record Dates: First submitted 2021-12-27; First posted 2022-01-27 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Locally Advanced Cervical Carcinoma
Keywords: Hypofractionation; Nodal simultaneous integrated boost; Intensity-modulated radiotherapy
MeSH Terms: interventions — Radiation Dose Hypofractionation; Brachytherapy

STUDY DESIGN:
Intervention Model Description: Two-phase study Phase 1: Dose-escalation study using standard 3+3 design Phase 2: Single-arm clinical trial using Simon's two-stage design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Hypofractionation — Phase 1 (Dose Escalation Study):
  Pelvic hypofractionated radiotherapy (40 Gy over 15 daily fractions) with nSIB 45 Gy (first dose level) and 48 Gy (second dose level); to be followed by brachytherapy (6.5-7.5 Gy x 4 fractions)
  Phase 2 (Efficacy Study):
  Pelvic hypofractionated radiotherapy (40 Gy over 15 daily fractions) with (or without) nSIB 45-48 Gy (depending on phase 1 results); to be followed by brachytherapy (6.5-7.5 Gy x 4 fractions)
  Other Names: Nodal simultaneous integrated boost; Brachytherapy

SUMMARY:
BACKGROUND: For patients with locally advanced cervical cancer (LACC) ineligible for concurrent chemotherapy, radiotherapy (RT) alone achieves complete response rate (CRR) <70% and long-term locoregional control (LRC) <62%. Hypofractionated (HF-)RT using older techniques results in comparable CRR and disease control, and low late toxicity rates (4-8%). Dose-adapted HF-RT using intensity-modulated radiotherapy (IMRT) with nodal simultaneous integrated boost (nSIB) could improve tumor control and toxicity.

GENERAL OBJECTIVE: To determine the effectiveness and safety of HF-RT with (or without) nSIB in LACC among patients who are chemo-ineligible.

PRIMARY OBJECTIVES:

Phase 1: To determine the maximum tolerated dose (MTD) for nSIB used in combination with pelvic HF-RT (2.67 Gray (Gy) x 15 fractions), using IMRT Phase 2: To assess the efficacy of HF-RT ± nSIB in terms of complete response rates at 3 months

SECONDARY OBJECTIVES:

To assess the efficacy of HF-RT ± nSIB in terms of progression free survival (PFS), locoregional PFS, distant metastasis free survival (DMFS), cervical cancer specific survival (CCSS), overall survival (OS)

To assess the acute and late toxicity of HF-RT ± nSIB, and patient-reported quality of life outcomes

EXPLORATORY OBJECTIVES:

To evaluate the predictive utility of clinical and dosimetric variables for tumor response/control and toxicity. Variables: age, performance status, T- and N-stage, T-score, histology, baseline hemoglobin, clinical target volume and organs-at-risk doses, overall treatment time

STUDY DESIGN:

Phase 1: Dose-escalation study (standard 3+3 design) Phase 2: Single-arm clinical trial (Simon's two-stage design)

STUDY TREATMENTS:

Pelvic HF-RT ± nSIB to 40 Gy in 15 fractions using IMRT, followed by brachytherapy (BRT) 6.5-7.5 Gy x 4 fractions using 2D or image-guided techniques

SAMPLE SIZE:

One-sided hypothesis testing. H0: CRR p0 ≤64%; H1: CRR p1 ≥84%. Simon 2 stage: First stage, n1=28 will be enrolled. If response (r1) ≤18, the study will be stopped for futility. Otherwise, second stage: n2=22, for a total of 50.

H0 will be rejected if r1+r2 ≥38, in 50 patients. This yields a type I error rate of 5% and power of 95% when the true response rate is ≥84%.

Accrual: Accounting for 10% attrition, a n=55 will be targeted. At a rate of 4-5 patients quarterly, accrual may take 33-42 months. The trial may be opened to other centers to accelerate accrual.

DETAILED DESCRIPTION:
SAMPLE SIZE CALCULATION:

CRR with chemoradiotherapy based on a meta-analysis in 2017 is about 80%; with advanced RT techniques, based on a multi-center, prospective study, local control rate >90% could be achieved.

Based on retrospective studies, CRR with HF-RT without concurrent chemotherapy (ChT) followed by BRT, using 2D techniques, is about 70%. This is comparable to CRR for conventionally fractionated RT without concurrent ChT in the above meta-analysis. Given the retrospective nature of HF-RT data, a low CRR of 64% could be projected (p0). Given that in the current study, the investigators propose to do dose-adapted radiation by using more advanced RT and BRT, a high CRR of 84% could be projected (p1).

In the first stage, 28 patients will be accrued, including the 3 or 6 patients enrolled in the MTD level from phase 1. If there are ≤18 responses in these 28 patients, the study will be stopped. Otherwise, 22 additional patients will be accrued in the second stage, for a total of 50.

The null hypothesis will be rejected if >38 responses are observed in 50 patients. This design yields a type I error rate of 5% and power of 95% when the true response rate is ≥84%.

Accounting for 10% attrition, a sample size of 55 will be targeted.

INDICATION:

Patients must meet all the inclusion criteria and none of the exclusion criteria to be eligible for this trial. Contraindication to ChT may be due to a medical contraindication or patient refusal to receive chemotherapy, and will be documented by the referring/attending gynecologic oncologist in the referral letter.

To effectively manage any conflict of interest, the attending/referring gynecologic oncologist shall not participate in the recruitment process. Any eligible patient will be referred to the Radiation Oncology Department, where the recruitment process will be initiated by the Primary Investigator or a delegated radiation oncology consultant.

TREATMENT REGIMEN:

The regimen consists of whole pelvic photon RT, using IMRT, followed by high dose rate (HDR) BRT. Inguinal fields shall be included in case of lower vaginal or inguinal nodal involvement. The prescription dose is 40 Gy in 15 fractions at 2.67 Gy/fraction.

The nSIB in the phase 2 will be given according to the MTD level in phase 1. The nSIB is indicated for any adenopathy detected by either positron emission tomography (PET)-positivity, by computed tomography (CT)/ magnetic resonance imaging (MRI) criteria such as a short axis diameter >10mm (15mm, for inguinal nodes), or histologically positive on surgical sampling. The gross nodal planning target volume (PTV) boost will receive 45-48 Gy in 3.0-3.2 Gy/fraction, depending on the projected contribution of BRT and location of the lymph node. Assuming both nodal boost dose levels are found to be associated with acceptable toxicity: common iliac or inguinal nodes will be boosted to 48 Gy; and external or internal iliac nodes, to 45 Gy given the BRT contribution to the total nodal dose.

The RT will be given once daily from Monday to Friday, 5 fractions per week.

BRT will be given after completion of pelvic RT, ideally within two weeks from completion. Two insertions per week may be done. If multiple fractions will be given using the same implant, these will be given twice daily, 6 hours apart.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged ≥18 years
2. Histologically confirmed cervical squamous, adeno-, or adenosquamous carcinoma
3. 2018 Fédération Internationale de Gynécologie et d'Obstétrique (FIGO) Stage IIIA-IIIC1, IVA
4. Pelvic nodal metastases (for the phase 1 cohorts)
5. Contraindication to chemotherapy
6. Brachytherapy candidate
7. World Health Organization (WHO)/ECOG performance status of ≤2
8. Life expectancy of at least 12 weeks
9. Adequate bone marrow function: Absolute neutrophil count ≥1,500 cell/mm3; Platelets ≥100,000 cell/mm3; Hemoglobin ≥10.0 g/dL; Leukocyte count ≥4,000 cell/mm3

Exclusion Criteria:

1. Other histology (small cell, neuroendocrine, lymphoma, sarcoma, etc.)
2. 2018 FIGO Stage IIIC2 (para-aortic nodal metastases)
3. Clinical and/or radiologic evidence of metastatic disease
4. History of another malignancy except for the following: malignancy treated with curative intent and with no known active disease ≥5 years and of low potential risk for recurrence; adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; adequately treated carcinoma-in-situ without evidence of disease
5. Pregnancy
6. Uncontrolled concurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, active interstitial lung disease, serious chronic GI conditions associated with diarrhea (including Crohn's disease or ulcerative colitis), or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events or compromise the ability of the patient to give written informed consent
7. Presence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule, including alcohol dependence or drug abuse
8. Prior hysterectomy
9. Prior treatment for cervical cancer
10. Prior pelvic radiotherapy
11. Concomitant anti-cancer therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (for phase 1) | 4 months
  The highest dose studied for which the incidence of dose-limiting toxicity was less than 33%
Complete response rate (for phase 2) | 3 months
  Proportion of treated patients with disappearance of all lesions on clinical and radiologic examination

SECONDARY OUTCOMES:
Progression-free survival | 5 years
  Time from date of enrolment to date of progression, date of death from any cause, or date of last follow-up, whichever occurs first
Locoregional progression-free survival | 5 years
  Time from date of enrolment to date of locoregional progression, date of death from any cause, or date of last follow-up, whichever occurs first
Metastasis-free survival | 5 years
  Time from date of enrolment to date of development of metastasis, date of death from any cause, or date of last follow-up, whichever occurs first
Cervical cancer-specific survival | 5 years
  Time from date of enrolment to date of death attributed to cervical cancer, or date of last-follow-up, whichever occurs first
Overall survival | 5 years
  Time from date of enrolment to date of death from any cause, or date of last follow-up, whichever occurs first
Acute and subacute toxicity | 4 months
  Radiation toxicity per RTOG criteria documented during and within 3-4 months from completion of treatment
Late toxicity | 5 years
  Radiation toxicity per RTOG criteria documented beyond 4 months from completion of treatment
Expanded Prostate Index Composite - Urinary Domain Scores | 5 years
  Multi-item questionnaire on urinary function, with scores transformed linearly from 0-100, with higher scores representing better quality of life.
Expanded Prostate Index Composite - Bowel Domain Scores | 5 years
  Multi-item questionnaire on bowel function, with scores transformed linearly from 0-100, with higher scores representing better quality of life.
European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core 30 Scores | 5 years
  Multi-item questionnaire on functions, symptoms and global quality of life, with scores transformed linearly from 0-100, with higher scores representing better quality of life.
European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Cervix 24 Scores | 5 years
  Multi-item questionnaire on cervical cancer specific aspects of quality of life, with scores transformed linearly from 0-100, with higher scores representing better quality of life.
Patient's Global Impression of Change (PGIC) | 5 years
  Reflects a patient's belief about the efficacy of treatment, from 1-7, with higher scores representing better patient's rating of overall improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bacorro, MD, Principal Investigator — University of Santo Tomas Hospital, Philippines

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data by emailing the primary investigator. All request will be evaluated by the study team and the USTH-REC.
Supporting Information: Study Protocol, SAP
Time Frame: Six months after publication
Access Criteria: When a request has been approved the study team will provide access to the de-identified individual patient-level data. Signed Data Sharing Agreement must be in place before accessing requested information. Additionally, all users will need to accept specified terms and conditions to gain access.

REFERENCES:
- [Background] Bacorro W, Baldivia K, Dumago M, Bojador M, Milo A, Trinidad CM, Mariano J, Gonzalez G, Sy Ortin T. Phase 1/2 trial evaluating the effectiveness and safety of dose-adapted Hypofractionated pelvic radiotherapy for Advanced Cervical cancers INeligible for ChemoTherapy (HYACINCT). Acta Oncol. 2022 Jun;61(6):688-697. doi: 10.1080/0284186X.2022.2048070. Epub 2022 Mar 14. PMID 35285405